CLINICAL TRIAL: NCT02815072
Title: Generation of Marfan Syndrome and Fontan Cardiovascular Models Using Patient-specific Induced Pluripotent Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/596/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-01

CONDITIONS: Marfan's Syndrome
Keywords: Fontan palliation; Marfan's syndrome
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 tablespoons of blood (20ml) will be taken for pre screening
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Skin biopsy — A sample of skin (approximately 0.5cm x 0.5cm) from inner thigh area. The skin biopsy will be conducted and completed with a single stitch to close the wound under local anaesthesia to minimise any discomfort. The skin biopsy will be taken by the medical doctor trained in biopsy collection. The tissue sample will be processed and cells will be grown out of them under appropriate conditions. These cells will only be used for laboratory experiments that include experimental transplantation models and laboratory bench-top research.

SUMMARY:
Medical researchers of National Heart Centre Singapore will carry out a state-of-the-art study that examines the possibility of changing patients' own cells into multi-functional and potent stem cells called iPS cells. These iPS cells can subsequently give rise to functional cardiac cells (myocytes) and other cardiovascular cells which might give further clues into the manifestation of the structural heart disease. This study involves blood sample collection for pre-screening and skin biopsies to establish skin cell culture.

DETAILED DESCRIPTION:
Participants are invited to participate in this study because they have been diagnosed with Marfan's syndrome whereby a gene mutation is suspected to have affected major blood vessel of their heart or have a Fontan procedure that was carried out to re-direct blood flow in their heart. This study will recruit 30 subjects from National Heart Centre Singapore over a period of 1 year.

For clinically diagnosed Marfan disease, a genetic test in a gene called FBN1 will be carried out to confirm the presence of gene mutation that is suspected to cause the disease. It is important for them to know that any research finding that indicates the presence of this gene mutation may only suggest a pre-disposition to Marfan disease, but it does not definitely ascertain that gene has caused the disease or predict that they will develop the disease. Further independent clinical genetic testing may be made available, should they so desire after consulting their doctor or genetic counsellor.

The skin obtained during the course of this study will be used for this study only and will be stored and analysed for the purposes of this study only, for a period not exceeding 5 years for research studies and experimental transplant studies, and will be destroyed after completion of the study, unless they agree to donate the samples to National Heart Centre Singapore for continuous storage for future studies that are approved by Institutional review board. The blood will however be stored indefinitely in National Heart Centre for future research on molecular, imaging and outcome studies of cardiovascular health and disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient that are under the care of the cardiologist and diagnosed with Marfan's syndrome or who had underwent Fontan palliation

Exclusion Criteria:

* No

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants who have been diagnosed with Marfan's syndrome whereby a gene mutation is suspected to have affected major blood vessel of their heart or have a Fontan procedure that was carried out to re-direct blood flow in their heart.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Generation of Marfan Syndrome and Fontan Cardiovascular Models using Patient-specific Induced Pluripotent Stem Cells | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ju Le Tan, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooke BS, Habashi JP, Judge DP, Patel N, Loeys B, Dietz HC 3rd. Angiotensin II blockade and aortic-root dilation in Marfan's syndrome. N Engl J Med. 2008 Jun 26;358(26):2787-95. doi: 10.1056/NEJMoa0706585. PMID 18579813
- [Background] Jin SM, Noh CI, Bae EJ, Choi JY, Yun YS. Impaired vascular function in patients with Fontan circulation. Int J Cardiol. 2007 Aug 21;120(2):221-6. doi: 10.1016/j.ijcard.2006.09.020. Epub 2006 Dec 18. PMID 17175041